CLINICAL TRIAL: NCT04672876
Title: Telotristat Ethyl for Reducing the Incidence of Intraoperative Carcinoid Crisis in Patients With Small Bowel Neuroendocrine Tumors
Brief Title: Telotristat Ethyl for Reducing Intraoperative Carcinoid Crisis in Patients With Neuroendocrine Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial funding no longer available.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0207
Record Dates: First submitted 2020-09-29; First posted 2020-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumors; carcinoid crisis; carcinoid tumors; surgery for carcinoid tumor; telotristat ethyl
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor | interventions — telotristat ethyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Telotristat Ethyl (Xermelo®) (Experimental): After the surgery is performed, study participants will stop taking telotristat ethyl (Xermelo®) as part of this study and there will be no follow-up visits or calls required outside of the usual postoperative care. The research team will collect clinical data on the participants' outcomes up to 30 days after surgery by accessing medical records.
  Interventions: Drug: Telotristat Ethyl Oral Tablet

INTERVENTIONS:
Drug: Telotristat Ethyl Oral Tablet — XERMELO is a prescription pill, used along with somatostatin analog (SSA) therapy, for Carcinoid Syndrome diarrhea in adults who are not adequately controlled by SSA therapy. The drug is currently FDA-approved for this use but this study has received special approval from the FDA (under an Investigational Drug Application) to study telotristat ethyl in individuals with carcinoid tumors who plan to undergo surgery.
  Other Names: Xermelo

SUMMARY:
This is a study to determine if a certain drug, called telotristat ethyl (Xermelo®), can help reduce the chance of blood pressure and heart rate variations (known as carcinoid crisis) in individuals who have neuroendocrine tumors (also called carcinoid tumors). These complications can be life-threatening for patients who already have to experience challenging surgeries to remove their tumors. To determine if telotristat ethyl (Xermelo®) will help reduce these complications during surgery, researchers will give the drug to study participants before surgery.

DETAILED DESCRIPTION:
What is carcinoid crisis and why study telotristat ethyl to help reduce it? Surgery and anesthesia can cause sudden, dangerous, difficult-to-control changes in blood pressure and heart rate (a "carcinoid crisis") in patients with carcinoid tumors. Patients who have crises for a duration of 10 minutes or longer have a 12-fold increased risk of major complications during surgery.

Historically, it has been believed that crises were due to a massive release of carcinoid hormones from tumors in the blood; therefore, this study will investigate if telotristat ethyl (Xermelo®) can help block this hormone release and reduce the rate of dangerous complications that patients with carcinoid tumors may experience during surgery to remove their tumors.

What will this study involve and how long will it last for participants? The study involves blood tests before, during and after surgery, and taking telotristat ethyl (Xermelo®) tablets orally for two weeks before surgery and on the day of surgery (no later than 2 hours prior to surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a grade 1 or grade 2 small bowel, neuroendocrine tumor (NET) that has been medically confirmed by a physician.
* Patients who plan to have abdominal (stomach) surgery due to cancer that has spread to their liver. Patients must voluntarily choose to have surgery.
* 18 years old or older.
* Patients with small bowel neuroendocrine tumors who are asymptomatic (not showing symptoms) but have elevated serotonin or 5-HIAA (5-hydroxyindoleacetic acid) levels before surgery.
* Patients who are symptomatic (showing carcinoid symptoms) and have elevated or normal Serotonin or 5-HIAA levels (plasma or urinary) before surgery.

Exclusion Criteria:

* Patients belonging to vulnerable populations such as children and prisoners.
* Patients with grade 3 neuroendocrine tumors or neuroendocrine tumors that are hard to identify.
* Patients with untreated carcinoid heart disease.
* Patients who are receiving any other drugs or treatment as part of a research study.
* Patients with a "currently active" second tumor other than non-melanoma skin cancers. Patients are not considered to have a "currently active" tumor if they have completed therapy and are free of disease for 3 or more years.
* Patients with known brain cancers.
* Patients who have a history of allergic reactions to medications that have similar chemical or biologic ingredients as those found in telotristat ethyl.
* Uncontrolled illness that occurs while having cancer such as, but not limited to, ongoing or active infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit the patient's ability to follow study requirements.
* Pregnant women are excluded from this study because telotristat ethyl can severely damage an embryo/fetus or cause an abortion. Because the drug also poses unknown, potential risks for nursing infants, breastfeeding should be discontinued if the mother is treated with telotristat ethyl.
* Women of childbearing age who refuse to take a urinary pregnancy test and refuse to use an acceptable method of birth control during the time of the study and for at least 7 days after surgery. Acceptable contraception includes barrier method (male or female condom); hormonal (oral or implantable); documented sterilization procedure; cap, diaphragm, or sponge with spermicide; or abstinence as a lifestyle choice.
* Patients on CYP3A4 substrates that cannot be stopped due to medical concerns for 15 days prior to surgery.
* Patients with moderate or severe liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Observed Carcinoid Crises During Surgery | 15 days (including day of surgery).
  To determine if surgical treatment with telotristat ethyl reduces the incidence of carcinoid crisis during surgery for participants with small bowel neuroendocrine tumors by comparing data from this study to data from previous research.